CLINICAL TRIAL: NCT04869254
Title: Correlation Between the Pre-transplantation Lymphocyte Count, Administered Dose of Thymoglobulin and Graft Versus Host Disease (GVHD) in Pediatric Recipients of Hematopoietic Stem Cells Transplantation: a Retrospective Study
Brief Title: Lymphocyte Count, ATG Dose and Incidence and Severity of GVHD in Pediatric Recipients of HSCT
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 08/2019
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Gvhd prophylaxis; pediatric patients; hematopoietic cell transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematopoietic stem cells transplantation: patients undergone allogeneic or autologous bone marrow transplant who received immunomodulatory therapy with Thymoglobulin
  Interventions: Other: Lower lymphocyte/ATG ratio; Other: Higher lymphocyte/ATG ratio

INTERVENTIONS:
Other: Lower lymphocyte/ATG ratio
  Other Names: Lymphocyte/ATG ratio <0.01
Other: Higher lymphocyte/ATG ratio
  Other Names: Lymphocyte/ATG ratio >0.01

SUMMARY:
Despite increasing success rate in hematopoietic stem cell transplantation (HSCT) control of graft versus host disease (GVHD) remains a significative burden in mortality and morbidity. A lot of strategies could lower the incidence and gravity of the disease and immunosuppressive treatment as GVHD prophylaxis still represent the main method.

Although immunosuppressive treatment showed a good effect on GVHD mortality a lot of studies also highlight an increase of relapse and infection related mortality that jeopardize the effect on overall survival of HSCT recipient. Using anti thymocyte globulin (ATG) as GVHD prophylaxis shares the same double-edge effect as other immunosuppressive treatment although is still unclear how manage dose and timing of the infusion to minimize promoting effect on infections and maximize protective effect on GVHD. Biological effect of ATG lead to a dose- related delay in all class of T-cell reconstitution but our data are mostly from adult studies with high doses between 30 and 60 mg/kg due to the more important burden of GVHD in HSCT adult population. As for other treatment in HSCT conditioning we would like to study a personalized approach for ATG treatment: some studies focus on tuning of ATG dose for kilos but previous evidence showed that the same dose could made too little or too much immunosuppressive effect for different patients, even though same age and same stem cell source.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the patients between 0 and 17
2. Diagnosis of hematological or oncological disease undergoing allogeneic bone marrow transplantation
3. Patients undergoing myeloablative conditioning
4. Patients that received ATG as GVHD prophylaxis
5. Patients whose consent has already been acquired for the processing of data for research purposes
6. Minimum follow-up of 12 months

Exclusion Criteria:

1. Bacterial and / or fungal infection present at the time of bone marrow transplantation
2. Use of Thymoglobulin in the 3 months prior to transplantation
3. Allergy and / or intolerance to the active substances or excipients contained in Thymoglobulin

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric recipients of hematopoietic stem cells transplantation
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Development of GVHD according to lymphocyte/ATG ratio | 24 months after transplant
  Differences in the frequency of GVHD according to the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01). Adjustment for potentially associated variables (e.g., dose of drug actually received by patients, age of patients, type of conditioning, underlying disease, type of donor) will be carried out

SECONDARY OUTCOMES:
Transplant related mortality according to lymphocyte/ATG ratio | 24 months after transplant
  Comparison of transplant related mortality 24 months after HSCT in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)
Incidence of Graft Failure according to lymphocyte/ATG ratio | 24 months after transplant
  Frequency of engraftment failure and hematological reconstitution time (defined as the first post-transplant day of at least three consecutive days with the presence of at least 500 neutrophils / mmc for myeloid engraftment and the first appearance of lymphoid cell subpopulations) in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)
Number of episodes of sepsis during the post-transplant period according to lymphocyte/ATG ratio | 24 months after transplant
  Number of episodes of sepsis after HSCT and correlated mortality and morbidity in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)
Number of episodes of fungal infections during the post transplant period according to lymphocyte/ATG ratio | 24 months after transplant
  Number of episodes of fungal infections after HSCT and correlated mortality and morbidity in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)
Number of episodes of viral reactivations during the post transplant period according to lymphocyte/ATG ratio | 24 months after transplant
  Number of episodes of viral reactivations after HSCT and correlated mortality and morbidity in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)
Entity of GVHD according to lymphocyte/ATG ratio | 24 months after transplant
  Severity and organ involvement of acute and chronic GVHD defined by the Glucksberg classification by degrees of severity in the two exposure's groups (lymphocyte/ATG ratio <0.01 vs >0.01)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Study Chair — IRCCS Burlo Garofolo; Alessandra Maestro, PharmD PhD, Study Director — IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided